CLINICAL TRIAL: NCT00866073
Title: Phase II Study of Low-Dose Intravenous Decitabine in Patients Aged > 60 Years With Acute Myeloid Leukemia Who Are Not Eligible for Standard Induction Chemotherapy
Brief Title: Study of Low-Dose Intravenous Decitabine in Patients Aged > 60 Years With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Prof. Dr. med. M. Lübbert, Dept. of Oncology/Hematology - University Medical Center Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00331
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Acute myeloid leukemia; Decitabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Decitabine 15 mg/m2 i.v. - single arm
  Interventions: Drug: Decitabine 15 mg/m2 i.v.

INTERVENTIONS:
Drug: Decitabine 15 mg/m2 i.v. — Decitabine at 15 mg/m2 i.v. x 3 hours, three times daily on three consecutive days
  Other Names: Dacogen

SUMMARY:
This study is an open-label phase II trial to investigate the efficacy and toxicity of low-dose decitabine (5-aza-2'-deoxycytidine) in elderly patients with acute myeloid leukemia (AML) not eligible for aggressive induction chemotherapy. AML patients above the age of 60 years (no upper age limit) who have not previously received and are not eligible for, standard induction treatment of their disease will be eligible for this trial. Decitabine will be administered as a 3 hour infusion at 15 mg/m2 three times daily on three consecutive days (total dose 135 mg/m2). In all patients with > 20000 WBC/µl, this treatment will be repeated 1 week later. In patients with white blood cells exceeding 50 000/μl, decitabine treatment will be preceded by cytoreductive doses of hydroxyurea.

DETAILED DESCRIPTION:
Hypothesis: If after 4 courses of Decitabine none out of 12 patients achieves a response (complete or partial remission, antileukemic effect), the protocol will be stopped. If at least one response is seen among the first 12 patients, 17 additional patients will be treated in an open, uncontrolled manner. If in 3 or more of these 29 patients a response is achieved, this treatment will be considered effective and will be studied further, otherwise it will be considered ineffective. At a preliminary analysis after recruitment of 29 patients, encouraging results (response rate, tolerability) are prompting continuation of recruitment, with a planned inclusion of at least 60 patients, until initiation of the planned large, controlled phase II follow-up trial. Unexpected toxicities will be carefully evaluated. 29 patients were needed for the first two steps of this phase II study, at least 60 patients are planned for the extension of the recruitment. Expected study duration for the first two steps was 15-20 months, with 35-40 months total when including the third step.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 60 years with acute myeloid leukemia (> 30 % bone marrow blasts) not qualifying for, or not consenting to, standard induction chemotherapy or immediate allografting
* life expectancy > 3 months with successful treatment
* performance status ECOG 0, 1, 2
* age-adjusted normal cardiac, kidney, liver function (creatinine < 1.5 mg/dl unless leukemia-related, total bilirubin < 2.0 of upper normal limits)
* patients with >50 000 leukocytes/µl in whom initial cytoreduction according to protocol is effective
* written informed consent

Exclusion Criteria:

* AML of FAB subtype M3
* previous induction-type chemotherapy for MDS or AML
* previous treatment with Decitabine, 5-azacytidine or ATRA
* "low-dose" chemotherapy (e.g.hydroxyurea, cytosine arabinoside, melphalan) within 8 weeks prior to Decitabine treatment, except for cytoreduction of leukocytosis > 50 000/µl according to protocol - patients with > 50 000 leukocytes/µl in whom initial cytoreduction according to protocol is ineffective
* treatment with cytokines within previous 4 weeks
* concomitant use of any other investigational drug
* other malignancy that is not in remission (previous chemotherapy for other malignancies is not an exclusion criteria)
* cardiac insufficiency NYHA IV
* HIV infection
* other uncontrolled active infection
* psychiatric disorder that interferes with treatment
* known hypersensitivity to retinoids
* contact lenses

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2003-04; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
response rate (complete and partial remissions, antileukemic effect) | after four treatment courses of Decitabine, after 6 months

SECONDARY OUTCOMES:
overall survival | after 1 year
progression-free survival time | after 1 year
toxicity of Decitabine (alone and in combination with all-trans retinoic acid) | after 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lübbert, Prof Dr med, Principal Investigator — University Medical Center Freiburg - Dept. of Oncology/Hematoloy
Locations (8):
- Germany (7):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Klinikum der Technischen Universität Aachen, Aachen
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Katholisches Krankenhaus Hagen, Hagen
  - Klinikum Lüdenscheid, Lüdenscheid
  - Universitätsklinikum Ulm, Ulm
  - Klinikum Villingen-Schwenningen, Villingen-Schwenningen
- Leyenburg Hospital, The Hague, Netherlands